CLINICAL TRIAL: NCT00566358
Title: Lightening the Hormonal Mechanisms of Surgical Treatment of Type 2 Diabetes Mellitus by Duodenal Exclusion Surgery
Brief Title: Surgical Treatment of Non-obese Type 2 Diabetic Patients With Duodenal Exclusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Bruno Geloneze, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIMED0002
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus, type 2; duodenal exclusion; bariatric surgery; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; insulin; glucagon; ghrelin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Duodenal exclusion
  Interventions: Procedure: Duodenal exclusion surgery

INTERVENTIONS:
Procedure: Duodenal exclusion surgery — Under open laparotomy, a duodenum section 2cm below the pylorus and a jejunum section below Treitz's Angle to create an excluded biliopancreatic limb of 150cm. A Roux-in-Y retrocolic anastomosis of the alimentary limb promotes the gastrojejunal continuity and the anastomosis of the excluded biliopancreatic limb is done 100cm below the jejunal-pyloric union.
  Other Names: Duodeno-jejunal exclusion; Duodenal-jejunal bypass

SUMMARY:
Diabetes reversion is observed after bariatric surgeries even before significant weight loss could explain it, mainly in predominantly malabsorptive procedures (98,9% for biliopancreatic diversion or duodenal switch), followed by those combining malabsorption and gastric restriction (83,7% for Roux-en-Y gastric bypass). Changes in the hormonal communication between the digestive system and the pancreas would explain the antidiabetogenic role of the surgery, so this effect could be obtained in nonobese, diabetic individuals.

In order to try this hypothesis, RUBINO and MARESCAUX (2004) studied the gastrojejunal bypass (duodenal exclusion)in an mouse model of diabetes without obesity. In their technique the stomach volume is kept intact, maintaining the caloric ingestion and the weight of the animals. There was a fast improvement of diabetes, independent of diet and weight, without the potential nutritional deprivations commonly seen in the bariatric surgery like iron and vitamin deficiency.

This study will evaluate the mechanisms of amelioration of type 2 diabetes mellitus after duodenal exclusion surgery in human non-obese, diabetic volunteers and known insulin secretion capacity, by the method of standardized meal stimulus. It is expected to be secondary to changes in the gastrointestinal hormones that stimulate insulin secretion (incretins).

The knowledge about the clinical outcomes of this technique in humans and the description of the secretion pattern of gastrointestinal hormones after the surgery may contribute to the implementation of this surgery as a new therapeutic option for overweight (non-obese) diabetic patients.

DETAILED DESCRIPTION:
There is large recovery of insulin sensibility after bariatric surgery, as the patients get closer to ideal weight. Diabetes reversion is more frequent after predominantly malabsorptive procedures (98,9% for biliopancreatic diversion or duodenal switch), followed by those combining malabsorption and gastric restriction (83,7% for Roux-en-Y gastric bypass). Glycemia normalization occurs in an early phase of the postoperative period, even before significant weight loss could explain it. These techniques have in common a bypass of the duodenum and part of the jejunum. Many peptides are released in this segments that regulate pancreatic beta cells (insulin producers) either in physiological state or in diabetes. Anatomical-functional changes in the enteroinsular axis would explain the antidiabetogenic role of the surgery, so this effect could be obtained in nonobese, diabetic individuals.

In order to try this hypothesis, RUBINO and MARESCAUX (2004) studied the gastrojejunal bypass (duodenal exclusion)in Goto-Kakizaki mice (GK), the most used animal model of diabetes without obesity. In their technique the stomach volume is kept intact, maintaining the caloric ingestion and the weight of the animals. There was a fast improvement of diabetes, independent of diet and weight. The authors concluded that this procedure should be applied in humans for reversal of diabetes without the potential nutritional deprivations commonly seen in the bariatric surgery like iron and vitamin deficiency.

The amelioration of diabetes after bariatric surgery is related to the modulation of production of gastrointestinal hormones relevant to the insulin production (incretin effect).

This study will evaluate the mechanisms of amelioration of type 2 diabetes mellitus after duodenal exclusion surgery in human non-obese, diabetic volunteers and known insulin secretion capacity, by the method of standardized meal stimulus. It is expected to be secondary to changes in the gastrointestinal hormones that stimulate insulin secretion (incretins).

The knowledge about the clinical outcomes of this technique in humans and the description of the secretion pattern of gastrointestinal hormones after the surgery may contribute to the implementation of this surgery as a new therapeutic option for overweight (non-obese) diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 60 years.
* BMI between 25 and 29,9 kg/m².
* Weight variance less than 5% in the last 3 months.
* Previous diagnosis of diabetes type 2.
* Insulin requirement, alone or along with oral agents
* Capacity to understand the procedures of the study.
* To agree voluntarily to participate of the study, signing an informed consent.

Exclusion Criteria:

* Positive Anti-GAD antibodies
* Laboratorial signal of probable failure of insulin production, i. e., seric peptide C lesser than 1 ng/mL.
* History of hepatic disease like cirrhosis or chronic active hepatitis.
* Kidney dysfunction (creatinine > 1,4 mg/dl in women and > 1,5 mg/dl in men).
* Hepatic dysfunction: ALT and/or AST 3x above upper normal limit.
* Recent history of neoplasia (< 5 years).
* Use of oral or injectable corticosteroids for more than consecutive 14 days in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Improvement or reversal of type 2 diabetes mellitus | 7 days, 14 days, 21 days, 1 month, 2 months, 3 months, six months and one year.
Changes in the secretion pattern of incretins, insulin and glucagon after intervention, as measured by standardized mixed meal tolerance test | 2 months, 6 months and 1 year

SECONDARY OUTCOMES:
Changes in body weight and fat distribution after intervention | 1 month, 2 months, 3 months, 6 months and 1 year
Changes in seric free fatty acids and lipoproteins | one month, 2 months, 3 months, 6 months and 1 year
Regression of carotid intima-media thickness | 1 month, 3 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Geloneze, MD, PhD, Principal Investigator — University of Campinas (UNICAMP); José Carlos Pareja, MD, PhD, Principal Investigator — University of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP), Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Rubino F, Marescaux J. Effect of duodenal-jejunal exclusion in a non-obese animal model of type 2 diabetes: a new perspective for an old disease. Ann Surg. 2004 Jan;239(1):1-11. doi: 10.1097/01.sla.0000102989.54824.fc. PMID 14685093
- [Result] Geloneze B, Geloneze SR, Fiori C, Stabe C, Tambascia MA, Chaim EA, Astiarraga BD, Pareja JC. Surgery for nonobese type 2 diabetic patients: an interventional study with duodenal-jejunal exclusion. Obes Surg. 2009 Aug;19(8):1077-83. doi: 10.1007/s11695-009-9844-4. Epub 2009 May 12. PMID 19475464